CLINICAL TRIAL: NCT01822431
Title: A Comparison Between Pupillometry, Heart Rate Variability and Metaiodobenzylguanidine Scintigraphy for the Diagnosis of Early Diabetic Autonomic Neuropathy in Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Zantidis Anestis, MD, AHEPA University Hospital
Other Study IDs: A-Z0001
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Autonomic Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with type 1 diabetes mellitus: Metaiodobenzylguanidine scintigraphy, Autonomic function tests, Pupillometry, Holter monitoring
  Interventions: Radiation: metaiodobenzylguanidine scintigraphy
- Healthy controls: Autonomic function tests, Pupillometry, Holter monitoring

INTERVENTIONS:
Radiation: metaiodobenzylguanidine scintigraphy
  Groups: Patients with type 1 diabetes mellitus

SUMMARY:
This study will examine if one of the following methods: pupillometry, spectral analysis of heart rate variability and metaiodobenzylguanidine scintigraphy, is more capable to detect early diabetic autonomic neuropathy in patients with type 1 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus

Exclusion Criteria:

* Type 2 diabetes mellitus
* Severe cardiac autonomic neuropathy
* Medications other than insulin
* Ocular disease other than refractive eye disorders
* History of neurologic disease
* History of cardiovascular disease
* Thyroid disease
* Vitamin B insufficiency
* Other possible cause for autonomic failure

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients: outpatient diabetes clinic of AHEPA university hospital Controls: residents of Thessaloniki area
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
number of participants with abnormal results | 1 day (at time of examination)

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA hospital, First Propedeutic clinic of internal medicine, Thessaloniki, Thessaloniki, Greece